CLINICAL TRIAL: NCT01030640
Title: A Phase 1, Randomized, Double- Blind (Sponsor-Open), Placebo-Controlled Study To Examine The Density Of Intraepidermal Nerve Fibers After A Single Subcutaneous Administration Of Tanezumab In Healthy Volunteers
Brief Title: Study To Assess Changes In The Number Of Nerves In The Skin At The Site Where Where Tanezumab Is Injected
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091046
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Osteoarthritis Pain; Chronic Low Back Pain; Pain Due to Interstitial Cystitis
Keywords: intraepidermal nerve fiber density; IENF; tanezumab; subcutaneous; healthy volunteers
MeSH Terms: interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): formulation without active drug
  Interventions: Other: placebo
- tanezumab (Active Comparator)
  Interventions: Biological: tanezumab

INTERVENTIONS:
Other: placebo — single dose of the drug formulation
  Arms: placebo
Biological: tanezumab — single dose of the active drug tanezumab at a dose level of 20 mg
  Arms: tanezumab

SUMMARY:
Subcutaneous administration of tanezumab can result in changes in the number of nerves around the injection site in the thigh.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects only
* Female subjects can not be pregnant or be nursing.
* Females and males need to use two types of birth control methods during the length of the study and one of the two methods needs to be a barrier method.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Subject can not have any chronic or acute medical condition or have had any chronic illness in the past
* Can not have any problematic skin condition.
* Females can not have more than 7 alcoholic drinks per week and males can not have more than 14 alcoholic drinks per week

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To assess the change in intraepidermal nerve fiber (IENF) density in skin biopsies from proximal thigh and distal leg between baseline and postdose time points after a single SC injection of tanezumab 20 mg SC or placebo in healthy volunteers. | 16 weeks
To compare the treatment effect between tanezumab 20 mg SC and placebo on the change in IENF density between baseline and postdose time points in skin biopsies from the proximal thigh and distal leg in healthy volunteers. | 16 weeks
To assess the safety, tolerability and immunogenicity of a single dose of tanezumab 20 mg SC in healthy volunteers. | 16 weeks

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of a single dose of tanezumab 20 mg SC administered in the proximal thigh in healthy volunteers | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091046&StudyName=Study%20To%20Assess%20Changes%20In%20The%20Number%20Of%20Nerves%20In%20The%20Skin%20At%20The%20Site%20Where%20Where%20Tanezumab%20Is%20Injected